CLINICAL TRIAL: NCT06891456
Title: Pulse Field Ablation for Post-Infarction Ventricular Tachycardia: the ASCEND Pilot Study
Brief Title: Pulsed Field Ablation for Post-Infarction Ventricular Tachycardia
Acronym: ASCEND-VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pasquale Santangeli (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Pasquale Santangeli, Sponsor-Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G250026
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Ventricular Tachycardia; Ischemic Heart Disease; Sustained VT
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- RFA Ablation (Active Comparator): VT ablation with ThermoCool ST, FlexAbility SE, ThermoCool ST SF or TactiFlex SE catheters
  Interventions: Device: RFA Ablation
- PFA Ablation (Experimental): VT ablation with FARAPOINT catheter
  Interventions: Device: PFA Ablation

INTERVENTIONS:
Device: RFA Ablation — RFA ablation of VT substrate using FlexAbility or ThermoCool ST catheter
  Arms: RFA Ablation
Device: PFA Ablation — PFA ablation of VT substrate using FARAPOINT catheter
  Arms: PFA Ablation

SUMMARY:
ASCEND is a randomized controlled open-label pilot study evaluating the safety and effectiveness of pulsed field ablation (PFA) with the novel FARAPOINT catheter compared to the standard radiofrequency (RFA) ablation with ThermoCool ST/FlexAbility SE/ThermoCool ST SF/TactiFlex SE of ventricular tachycardia (VT) in the patients with ischemic cardiomyopathy and implantable cardioverter-defibrillator (ICD). The study hypothesis is that the PFA ablation is more efficient compared to the RFA technique but retains a comparable safety profile.

DETAILED DESCRIPTION:
The ASCEND trial is a pilot study that will test the hypothesis that the novel FARAPOINT catheter and the FARAPULSE PFA platform can accomplish ischemic substrate VT ablation more efficiently and with a similar safety profile compared to a contemporary, widely adopted RFA technology (ThermoCool ST/FlexAbility SE/ThermoCool ST SF/TactiFlex SE).

ASCEND is a single center, controlled (two-arm), 1:1 parallel-randomized, open-label pilot study of 40 consecutively enrolled patients with ischemic cardiomyopathy and drug refractory or drug intolerant VT in whom a catheter ablation procedure is indicated. The study intervention consists of the use of a novel FARAPOINT PFA catheter during the entire VT ablation procedure. Patients randomized to the control arm of the study will undergo VT ablation using a contemporary standard-of-care technology (ThermoCool ST/FlexAbility SE/ThermoCool ST SF/TactiFlex SEcatheters).

This pilot study is designed to test for superiority with respect to the primary efficacy metric and to ensure comparable safety profiles of both ablation methods.

ELIGIBILITY:
Inclusion Criteria: must meet all of the following:

1. Age ≥18 years.
2. Ischemic heart disease with prior myocardial infarction.
3. Left ventricular ejection fraction ≥20% estimated by transthoracic echocardiography (TTE) within 90 days prior to enrollment.
4. Documented sustained monomorphic VT with any of the following characteristics:

   1. ≥2documented episodes in patients with implantable cardioverter defibrillators (ICD)
   2. ≥1 documented episode(s) in patients without ICD
   3. Recurrent VT despite antiarrhythmic medications (ineffective, contraindicated or not tolerated) or ICD interventions
5. Provision of signed and dated informed consent form.
6. Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria: any of the following:

1. Unable to provide informed consent.
2. Idiopathic VT.
3. Mobile LV thrombus.
4. Acute coronary syndrome within the preceding 2 months (if incessant VT ≥1 month before enrollment).
5. Comorbidity likely to limit survival to <12 months
6. New York Heart Association class IV heart failure.
7. Estimated glomerular filtration rate <30 ml/min/1.73m2.
8. Thrombocytopenia or coagulopathy.
9. Contraindication to heparin.
10. Pregnancy or lactation.
11. Cardiac surgery within the past 2 months.
12. Active infection.
13. Clinical, laboratory or imaging evidence of active ischemia.
14. Severe left heart valvular heart disease (aortic/mitral stenosis or regurgitation).
15. Any concomitant congenital heart disease.
16. Prior catheter or surgical ablation of VT within the past 2 months.
17. Anticipated need for epicardial mapping and ablation.
18. For individuals with no pre-existing ICD: Ineligibility for an ICD implant.
19. Pre-existing LVAD or other hemodynamic assist device
20. Present mechanical heart valve
21. cardiogenic shock unless it is due to incessant VT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedural Efficiency | Periprocedural
  Total ablation time (in seconds) needed to achieve complete elimination of late abnormal ventricular activities (LAVAs) in myocardial scar.
Procedural Safety | Within 7 days post procedure
  Count of individuals who experience any of the following:
  * Cardiac perforation
  * Pericardial effusion with hemodynamic compromise or needing intervention
  * New complete heart block
  * Coronary spasm
  * Acute MI
  * New acute severe mitral regurgitation or aortic regurgitation
  * Deep venous thrombosis
  * Vascular injury requiring surgical or percutaneous intervention
  * Pulmonary embolism
  * Stroke
  * Acute kidney injury
  * Death

SECONDARY OUTCOMES:
Secondary Safety | 180 days post procedure
  Changes in LVEF and/or new wall motion abnormalities at follow-up TTE

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Santangeli, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No